CLINICAL TRIAL: NCT00519636
Title: A Randomized, Double-blind, Placebo-controlled, Active Comparator, One-Week, Cross-Over, Multicenter Study to Evaluate the Efficacy and Patient Preference of Nasal Spray Characteristics of Once-Daily, Intranasal Administration of 110mcg Fluticasone Furoate Nasal Spray and 200mcg Fluticasone Propionate Nasal Spray in Adult Subjects With Seasonal Allergic Rhinitis
Brief Title: Comparator Study Evaluating Patient Experience And Preference Of FFNS vs. FPNS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FFU105927
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: experience; GW685698X; fluticasone furoate; preference; seasonal allergic rhinitis; fluticasone propionate
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal | interventions — Fluticasone; fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FFNS, FPNS (Active Comparator): fluticasone furoate nasal spray, fluticasone propionate nasal spray
  Interventions: Drug: FPNS; Drug: FFNS
- FPNS, FFNS (Active Comparator): fluticasone propionate nasal spray, fluticasone furoate nasal spray
  Interventions: Drug: FPNS; Drug: FFNS
- placebo FFNS, placebo FPNS (Placebo Comparator): placebo nasal spray matching fluticasone furoate nasal spray, placebo nasal spray matching fluticasone propionate nasal spray
  Interventions: Drug: placebo FFNS; Drug: placebo FPNS
- placebo FPNS, placebo FFNS (Placebo Comparator): placebo nasal spray matching fluticasone propionate nasal spray, placebo nasal spray matching fluticasone furoate nasal spray
  Interventions: Drug: placebo FFNS; Drug: placebo FPNS

INTERVENTIONS:
Drug: FPNS — fluticasone propionate nasal spray
  Other Names: fluticasone propionate; fluticasone furoate
  Arms: FFNS, FPNS; FPNS, FFNS
Drug: FFNS — fluticasone furoate nasal spray
  Arms: FFNS, FPNS; FPNS, FFNS
Drug: placebo FFNS — placebo nasal spray matching fluticasone furoate nasal spray
  Arms: placebo FFNS, placebo FPNS; placebo FPNS, placebo FFNS
Drug: placebo FPNS — placebo nasal spray matching fluticasone propionate nasal spray
  Arms: placebo FFNS, placebo FPNS; placebo FPNS, placebo FFNS

SUMMARY:
The purpose of this replicate study to FFU105924 is to provide data on subject preference of FFNS as compared with FPNS.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Active Comparator, One-Week, Cross-Over, Multicenter Study to Evaluate the Efficacy, Patient Preference and Experience of One-Daily, Intranasal Administration of 110mcg Fluticasone Furoate Nasal Spray and 200mcg Fluticasone Propionate Nasal Spray in Adult Subjects with Seasonal Allergic Rhinitis (FFU105927)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Subject has provided an appropriately signed and dated informed consent.
* Otherwise healthy outpatient with fall allergy
* Subject is treatable on an outpatient basis.
* Age
* 18 years or age or older at time of Visit 2
* Male or eligible female
* Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test will be required of all females at all visits to determine if the subject is pregnant.
* To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control, as defined by the following:
* Abstinence
* Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days).
* Oral contraceptive (either combined estrogen/progestin or progestin only)
* Injectable progestogen
* Implants of levonorgestrel
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year,
* Male partner who is sterile (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study and is the sole sexual partner for that female subject
* Double barrier method-condom or occlusive cap (diaphragm or cervical /vault caps) plus spermicide
* Estrogenic vaginal ring
* Diagnosis of SAR
* SAR is defined as follows:
* A clinical history (written or verbal) of SAR with seasonal allergy symptoms (nasal symptoms) during each of the last two fall allergy seasons, and
* A positive skin test (by prick method) to fall allergen prevalent to the geographic area during the conduct of the study, within 12 months prior to Visit 1 or at Visit 1.
* A positive skin test is defined as a wheal 3 mm larger than the diluent control for prick testing.
* In vitro tests for specific IgE (such as RAST, PRIST) will not be allowed as a diagnosis of SAR.
* Subjects who meet the above criteria and who may also have perennial allergic rhinitis or vasomotor rhinitis are eligible for randomization.
* Adequate exposure to seasonal pollen
* Subject resides within a geographical region where exposure to fall seasonal allergen is expected to be significant during the entire study period.
* Subject does not plan to travel outside this area for more than 48 hours of the study period.
* Ability to comply with study procedures
* Subject understands and is willing, able and likely to comply with study procedures and restrictions.
* Literate
* Subject must be able to read, comprehend, and record information in English.

Exclusion Criteria:

* Recent use (less than 1 year) of using branded (FLONASE) or generic FPNS or use of FFNS (VERAMYST).
* Significant concomitant medical conditions, defined as but not limited to:
* A historical or current evidence of clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.
* A severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation that could affect the deposition of intranasal study drug
* Nasal (eg, nasal septum) injury or surgery in the last 3 months
* Asthma, with the exception of mild intermittent asthma [National Asthma Education and Prevention Program (NARPP) Guidelines, 2002].
* Rhinitis medicamentosa
* Bacterial or viral infection (e.g., common cold) of the eyes or upper respiratory tract within two weeks of Visit 1 or during the screening period
* Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator
* Current or history of glaucoma and/or cataracts or ocular herpes simplex Physical impairment that would affect subject's ability to participate safely and fully in the study
* Clinical evidence of a Candida infection of the nose
* History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would confound the interpretation of the study results
* History of adrenal insufficiency
* History of shingles
* Chickenpox or measles: A subject is not eligible if he/she currently has chickenpox or measles, or has been exposed to chickenpox or measles during the last 3 weeks and is non-immune. If a subject develops chickenpox or measles during the study, he/she will be withdrawn from the study. If a non-immune subject is exposed to chickenpox or measles during the study, his/her continuation in the study will be at the discretion of the investigator, taking into consideration the likelihood of developing active disease.
* Use of other corticosteroids, defined as:
* Intranasal corticosteroid within four weeks prior to Visit 1.
* Inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less) within eight weeks prior to Visit 1.
* Use of other allergy medications within the timeframe indicated relative to Visit 1
* Intranasal cromolyn within 14 days prior to Visit 1
* Short-acting prescription and OTC antihistamines, including antihistamines contained in insomnia and 'nighttime' pain formulations taken for insomnia, within 3 days prior to Visit 1
* Long-acting antihistamines within 10 days prior to Visit 1: loratadine, desloratadine, fexofenadine, cetirizine
* Oral or intranasal decongestants within 3 days prior to Visit 1
* Intranasal, oral, or inhaled anticholinergics within 3 days prior to Visit 1
* Oral antileukotrienes within 3 days prior to Visit 1
* Subcutaneous omalizumab (Xolair) within 5 months of Visit 1
* Intranasal antihistamines (e.g. Astelin) within 2 weeks prior to Visit 1
* Use of other medications that may affect allergic rhinitis or its symptoms
* Chronic use of concomitant medications, such as tricyclic antidepressants, that would affect assessment of the effectiveness of the study drug
* Chronic use of long-acting beta-agonists (e.g., salmeterol)
* Chronic use of other intranasally administered medications (e.g., calcitonin-salmon)
* Nasal irrigation solutions
* Use of immunosuppressive medications 8 weeks prior to screening and during the study
* Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole
* Immunotherapy
* Subjects may be enrolled into the study if the immunotherapy was not initiated within 30 days of Visit 1, if the dose has remained fixed over the 30 days prior to Visit 1, and the dose will remain fixed for the duration of the study.
* Allergy/Intolerance
* Known hypersensitivity to corticosteroids or any excipients in the product
* Clinical trial/experimental medication experience
* Has recent exposure to an investigational study drug within 30 days of Visit 1
* Participation in a previous or current GSK FFNS study
* Positive or inconclusive pregnancy test or female who is breastfeeding
* Has a positive or inconclusive pregnancy test at Visit 1 or Visit 2
* Affiliation with investigational site
* Subject is a participating investigator, sub-investigator, study co-ordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.
* Current tobacco use
* Subject currently uses smoking products including cigarettes, cigars, and pipe or chewing tobacco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (23):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Rockville Centre, New York
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Meltzer EO, Andrews C, Journeay GE, Lim J, Prillaman BA, Garris C, Philpot E. Comparison of patient preference for sensory attributes of fluticasone furoate or fluticasone propionate in adults with seasonal allergic rhinitis: a randomized, placebo-controlled, double-blind study. Ann Allergy Asthma Immunol. 2010 Apr;104(4):331-8. doi: 10.1016/j.anai.2010.02.010. PMID 20408344
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFU105927 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone Furoate NS/Fluticasone Propionate NS: Subjects who received Fluticasone Furoate Nasal Spray(FFNS)110 mcg QD followed by Fluticasone Propionate Nasal Spray (FPNS) 200 mcg QD for one week(treatment 1), followed by a 7 day washout period, and switched to one week of treatment 2, given FPNS 110 mcg QD, followed by FFNS 200 mcg QD.
- Placebo FF/FP: Subject who received no active drug but believed they were following the Fluticasone Furoate/Fluticasone Propionate group.
- Fluticasone Propionate NS/Fluticasone Furoate NS: Subjects who received Fluticasone Propionate Nasal Spray (FPNS)110 mcg QD followed by Fluticasone Furoate Nasal Spray (FFNS) 200 mcg QD for one week(treatment 1), followed by a 7 day washout period, and switched to one week of treatment 2, given FFNS 110 mcg QD, followed by FPNS 200 mcg QD.
- Placebo FP/FF: Subjects who received no active drug but believed they were following the Fluticasone propionate/Fluticasone Furoate group.
Period: Treatment Period 1
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Started | 91 | 86 | 90 | 93
Completed | 89 | 86 | 89 | 93
Not Completed | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Sponsor request due to missed visit | 1 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Started | 89 | 86 | 89 | 93
Completed | 69 | 72 | 75 | 88
Not Completed | 20 | 14 | 14 | 5
Not completed — Adverse Event | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Failed to meet continuation criteria | 14 | 11 | 9 | 3
Not completed — Out of pollen area > 48 hours | 1 | 0 | 0 | 0
Not completed — Participating in study at another site | 1 | 0 | 0 | 0
Not completed — Non-compliant | 0 | 1 | 0 | 0
Not completed — Per doctors request | 0 | 1 | 0 | 0
Not completed — Subject randomized in error | 0 | 0 | 1 | 0
Not completed — Prohibited medications | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Started | 69 | 72 | 75 | 88
Completed | 69 | 71 | 74 | 86
Not Completed | 0 | 1 | 1 | 2
Not completed — Failed To Meet Continuation Criteria | 0 | 0 | 0 | 1
Not completed — Subject randomized in error | 0 | 1 | 0 | 0
Not completed — Per doctors request | 0 | 0 | 1 | 0
Not completed — Subject misrandomized | 0 | 0 | 0 | 1
Period: Post Study Period
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Started | 69 | 71 | 74 | 86
Completed | 69 | 71 | 74 | 85
Not Completed | 0 | 0 | 0 | 1
Not completed — Subject randomized in error | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF | Total
Number analyzed (Participants) | 91 | 86 | 90 | 93 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.25) | 38 (11.54) | 37.2 (12.55) | 38.9 (11.39) | 38.3 (11.91)
Gender [Count of Participants; unit: Participants]
  Female | 49 | 51 | 60 | 54 | 214
  Male | 42 | 35 | 30 | 39 | 146
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 15 | 11 | 23 | 21 | 70
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian: Central/South Asian Heritage | 1 | 2 | 1 | 3 | 7
  Asian: Japanese/East-Southeast Asian Heritage | 2 | 4 | 2 | 4 | 12
  Native Hawaiian or other Pacific Islander | 2 | 1 | 0 | 1 | 4
  White | 67 | 66 | 63 | 64 | 260
  African American/African Heritage & Asian | 1 | 0 | 0 | 0 | 1
  African American/African Heritage & White | 0 | 0 | 1 | 0 | 1
  Unknown | 2 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Mean Change From Baseline in Daily Reflective Total Nasal Symptom Score (rTNSS) Over Each Treatment Period of Active Drug Nasal Sprays Versus Placebos
Description: Reflective Total Nasal Symptom scores (rTNSS) symptoms of rhinorrhea, nasal congestion, nasal itching, sneezing using scale of: 0=none, 1=mild, 2=moderate, 3=severe; maximum score=12. The mean of AM and PM scores were used.
Time Frame: Baseline, Treatment Period 1 (Days 1-7), Treatment Period 2 (Days 15-21)
Population: Intent-to-Treat(ITT) population consisted of all subjects who were randomized to study treatment, and was to form the basis of all summaries of background, demographic, safety, and efficacy data.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Number analyzed (Participants) | 90 | 86 | 90 | 92
Scores on a scale
  Change from Baseline Treatment Period 1 | -2.7 (0.26) | -1.7 (0.22) | -2.2 (0.23) | -1.5 (0.22)
  Change from Baseline Treatment Period 2 | -2.7 (0.29) | -2.1 (0.27) | -2.3 (0.30) | -1.7 (0.26)
Statistical Analysis 1: Comparison: Fluticasone Furoate NS/Fluticasone Propionate NS vs Placebo FF/FP; FFNS combined across treatment arms 1 (FFNS/FPNS) & 2 (Placebo FF/FP) compared with Placebo FFNS combined across treatment arms 1 (FFNS/FPNS) & 2 (Placebo FF/FP); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.8, 95% CI [-1.3 to -0.3], Standard Error of Mean 0.24 — Mean Difference = Mean Change in FFNS - Mean Change in Placebo
Statistical Analysis 2: Comparison: Fluticasone Propionate NS/Fluticasone Furoate NS vs Placebo FP/FF; FPNS combined across treatment arms 1 (FPNS/FFNS) & 2 (Placebo FP/FF) compared with Placebo FPNS combined across treatment arms 1 (FPNS/FFNS)& 2 (Placebo FP/FF); Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Net) = -0.6, 95% CI [-1.1 to -0.1], Standard Error of Mean 0.24 — Mean Difference = Mean Change in FPNS - Mean Change in Placebo

2. Primary Outcome: Subject Preference of Fluticasone Furoate Nasal Spray (FFNS) Versus Fluticasone Propionate Nasal Spray (FPNS) Based on Scent/Odor
Description: Subjects assessed preference of scent/odor for the nasal sprays used during the treatment periods by answering "I prefer product 1" for spray used during Treatment Period 1 or "I prefer product 2" for spray used during Treatment Period 2. Subject could also choose "I have no preference."
Time Frame: End of Crossover Period (Day 22)
Population: Intent-to-Treat(ITT) population. These measures are from the product preference questionnaire given at the end of the study. Because questionnaires were comparative in nature, only subjects who completed both treatment periods were included in the analyses. In addition, there are small variations due to non-response for individual questions.
Measure: Number; unit: Participants
Groups:
- Total: All subjects on both arms preference.
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Fluticasone Propionate NS/Fluticasone Furoate NS | Total
Number analyzed (Participants) | 68 | 74 | 142
Participants
  Perferred - Fluticasone Furoate Nasal Spray | 41 | 41 | 82
  Perferred - Fluticasone Propionate Nasal Spray | 18 | 20 | 38
  No Preference | 9 | 13 | 22
Statistical Analysis 1: Comparison: Fluticasone Furoate NS/Fluticasone Propionate NS vs Fluticasone Propionate NS/Fluticasone Furoate NS; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel(CMH): stratified approximate to Prescotts test; variation of chi-square test for treatment sequence/subjects no preference

3. Secondary Outcome: Comparation of Mean Change From Baseline Over Each Treatment Period in Daytime Reflective Total Nasal Symptom Scores (D r-TNSS) for Active Drug Nasal Sprays Versus Placebos
Description: Reflective Total Nasal Symptom scores (rTNSS) symptoms of rhinorrhea, nasal congestion, nasal itching, sneezing using scale of: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: Baseline, Treatment Period 1 (Days 1-7), Treatment Period 2 (Days 15-21)
Population: Intent-to-Treat(ITT) population. A subject in the FP/FF group had no baseline daytime TNSS; however, does have a baseline nighttime TNSS, that value serves as the baseline 24-hour TNSS. Therefore there are 90 24-hour & nighttime TNSS observations available in the FP/FF group, but only 89 daytime TNSS observations.
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Placebo FF/FP: Subjects who received no active drug but believed they were following the Fluticasone Furoate/Fluticasone Propionate group.
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Number analyzed (Participants) | 90 | 86 | 89 | 92
Scores on a scale
  Change from Baseline- Treatment Period 1 | -2.9 (0.27) | -1.6 (0.22) | -2.4 (0.25) | -1.7 (0.23)
  Change from Baseline- Treatment Period 2 | -2.7 (0.29) | -2.2 (0.28) | -2.4 (0.32) | -1.9 (0.27)

4. Secondary Outcome: Comparision of Mean Change From Baseline Over Each Treatment Period in Nighttime Reflective Total Nasal Symptom Scores (N-rTNSS) for Active Drug Nasal Sprays Versus Placebos
Description: Reflective Total Nasal Symptom scores (rTNSS) symptoms of rhinorrhea, nasal congestion, nasal itching, sneezing using scale of: 0=none, 1=mild, 2=moderate, 3=severe; maximum score=12.
Time Frame: Baseline, Treatment Period 1 (Days 1-7), Treatment Period 2 (Days 15-21)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Placebo FF/FP | Fluticasone Propionate NS/Fluticasone Furoate NS | Placebo FP/FF
Number analyzed (Participants) | 90 | 86 | 90 | 92
Scores on a scale
  Change from Baseline- Treatment Period 1 | -2.7 (0.28) | -1.7 (0.23) | -2.1 (0.25) | -1.4 (0.24)
  Change from Baseline- Treatment Period 2 | -2.7 (0.32) | -2.0 (0.29) | -2.2 (0.32) | -1.6 (0.28)

5. Secondary Outcome: Subject Preference of Fluticasone Furoate Nasal Spray (FFNS) Versus Fluticasone Propionate Nasal Spray (FPNS) on Preference for: Leaking Out of Nose/Down Throat
Description: Subjects assessed preference over leaking out of nose/down throat for the nasal sprays used during the treatment periods by answering "I prefer product 1" for spray used during Treatment Period 1 or "I prefer product 2" for spray used during Treatment Period 2. Subject could also choose "I have no preference."
Time Frame: End of Crossover Period (Day 22)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Fluticasone Propionate NS/Fluticasone Furoate NS | Total
Number analyzed (Participants) | 69 | 73 | 142
Participants
  Preferred - Fluticasone Furoate Nasal Spray | 45 | 39 | 84
  Preferred - Fluticasone Propionate Nasal Spray | 16 | 14 | 30
  No Preference | 8 | 20 | 28

6. Secondary Outcome: Subject Preference of Fluticasone Furoate Nasal Spray (FFNS) Versus Fluticasone Propionate Nasal Spray (FPNS) on Preference for: Ease of Use
Description: Subjects assessed preference over ease of use for the nasal sprays used during the treatment periods by answering "I prefer product 1" for spray used during Treatment Period 1 or "I prefer product 2" for spray used during Treatment Period 2. Subject could also choose "I have no preference."
Time Frame: End of Crossover Period (Day 22)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Fluticasone Propionate NS/Fluticasone Furoate NS | Total
Number analyzed (Participants) | 69 | 74 | 143
Participants
  Preferred - Fluticasone Furoate Nasal Spray | 28 | 30 | 58
  Preferred - Fluticasone Propionate Nasal Spray | 22 | 32 | 54
  No Preference | 19 | 12 | 31

7. Secondary Outcome: Subject Preference of Fluticasone Furoate Nasal Spray (FFNS) Versus Fluticasone Propionate Nasal Spray (FPNS) on Preference for: Gentleness of Mist
Description: Subjects assessed preference over gentleness of mist for the nasal sprays used during the treatment periods by answering "I prefer product 1" for spray used during Treatment Period 1 or "I prefer product 2" for spray used during Treatment Period 2. Subject could also choose "I have no preference."
Time Frame: End of Crossover Period (Day 22)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fluticasone Furoate NS/Fluticasone Propionate NS | Fluticasone Propionate NS/Fluticasone Furoate NS | Total
Number analyzed (Participants) | 69 | 74 | 143
Participants
  Preferred - Fluticasone Furoate Nasal Spray | 38 | 44 | 82
  Preferred - Fluticasone Propionate Nasal Spray | 17 | 20 | 37
  No Preference | 14 | 10 | 24

ADVERSE EVENTS:
Description: Since this is a cross-over study, total number of participants reflect the total number per treatment per period.
Groups:
- Fluticasone Furoate Nasal Spray: Subjects who received Fluticasone Furoate.
- Fluticasone Propionate Nasal Spray: Subjects who receive Fluticasone Propionate Nasal Spray.
- Placebo - FF: Subjects who took no active drug but believed they were on Fluticasone Furoate Nasal Spray.
- Placebo -FP: Subject who took no active drug but believed they were on Fluticasone Propionate Nasal Spray.
Arm/Group | Fluticasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo - FF | Placebo -FP
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/159 | 0/174 | 0/166
Other Adverse Events (participants affected / at risk) | 7/166 | 14/159 | 12/174 | 12/166
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate Nasal Spray (N=166) | Fluticasone Propionate Nasal Spray (N=159) | Placebo - FF (N=174) | Placebo -FP (N=166)
Headache (Nervous system disorders) | 7 | 14 | 12 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.